CLINICAL TRIAL: NCT01749813
Title: Specific Carbohydrate Diet as Maintenance Therapy in Crohn's Disease
Acronym: SCD
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jennifer Burgis, Principle Investigator, Stanford University
Other Study IDs: 23031
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Crohn's Disease
Keywords: Carbohydrate Specific Diet; Crohn's Disease; Immunomodulators
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and stool
Oversight: Data Monitoring Committee: No

SUMMARY:
This study investigates whether the specific carbohydrate diet (SCD) can maintain clinical remission in pediatric and adult patients with Crohn's disease.

DETAILED DESCRIPTION:
Patients will be seen in clinic at new diagnosis of Crohn's disease or a flare of existing disease. Potential subjects will be screened with for eligibility, followed by a baseline assessment by the clinic provider. Subjects who wish to participate will undergo further discussion with one of the study staff. At enrollment, a member of the study staff will explain the study to the prospective participant (for consent and/or assent, if applicable given patient's age).

The SCD will be started in addition to previous maintenance medication therapy or with short course of corticosteroids 1-2mg/kg/day (up to 60mg maximum). Steroid induction based on clinical need.

We anticipate improvement in clinical symptoms, laboratory values and/or a decline in PCDAI of 12.5 points (pediatric patients) or decline in CDAI of 70 points (adult patients) after 4 weeks. Patients who do not reach remission by 4 weeks will be excluded from the study. Patients who require additional medications for disease control will be excluded from the study.

Patients will be seen in clinic at diagnosis, 2 weeks (if required by clinical symptoms), 1 month, 3 months and 6 months.

Assessment at initial enrollment and at all follow-up visits includes:

1. History of symptoms
2. Physical exam including height, weight, BMI, Tanner staging
3. Calculation of Pediatric Crohn's Disease Activity Index (PCDAI) for pediatric patients or the Crohn's Disease Activity Index (CDAI) score for adult patients.
4. Dietary assessment and nutritional counseling
5. Completion of validated quality of life measurement (IMPACT III for pediatric patients and SIBDQ in adult patients)
6. Adverse event monitoring (record of symptoms and review of laboratory surveillance)
7. Laboratory assessment including: CBC with differential, basic metabolic panel, liver function tests, albumin, ESR, CRP, stool calprotectin and stool lactoferrin
8. Serum sample for cytokine studies
9. Stool studies for microbiota studies

ELIGIBILITY:
Inclusion Criteria:

* Adult or pediatric patients presenting with a new diagnosis or flare of existing Crohn's disease based on standard diagnostic criteria including: clinical symptoms, laboratory parameters, disease activity indices (Pediatric Crohn's Disease Activity Index (PCDAI) for patients <19years and Crohn's Disease Activity Index (CDAI) for patients >19years), pathology from upper endoscopy/colonoscopy and imaging studies.

Exclusion Criteria:)

* Pregnancy
* Other autoimmune conditions including celiac disease, rheumatoid arthritis, multiple sclerosis
* Otherwise immunosuppressed patients including HIV and prior organ transplant
* Patients diagnosed with ulcerative colitis or indeterminate colitis
* Active tuberculosis

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children under 18 Adult
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2012-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Specific Carbohydrate Diet as Maintenance Therapy in Crohn's Disease | 1 year
  The primary end point of the study is the proportion of patients achieving steroid free remission at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ken Cox, MD, Principal Investigator — Stanford University Medical; Shamita Shah, MD, Principal Investigator — Stanford University Medicial; Jennifer Burgis, MD, Principal Investigator — Stanford University Medical
Locations (2):
- United States (2):
  - Stanford University Medical Center, Palo Alto, California
  - Stanford, Palo Alto, California

REFERENCES:
- See also: Specific Carbohydrate Diet in Crohn's Disease — http://med.stanford.edu/clinicaltrials/